CLINICAL TRIAL: NCT02222571
Title: Formative Research - Developing a Family-based Obesity Prevention Intervention in the Canadian Context
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Guelph (Other)
Collaborators: Danone Institute International (Other)
Responsible Party: Principal Investigator, Jess Haines, Assistant Professor, University of Guelph
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 12JL030
Record Dates: First submitted 2013-10-21; First posted 2014-08-21 (Estimated); Last update posted 2017-01-05 (Estimated); Status verified 2017-01

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Organization and Administration; Safety

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (Active Comparator): 9-week parenting group focused on safety
  Interventions: Behavioral: Supervision for Safety
- Parents and Tots Together Program (Experimental): Parents and Tots Together Program is a 9-week, group-based parenting intervention
  Interventions: Behavioral: Parents and Tots Together Program

INTERVENTIONS:
Behavioral: Parents and Tots Together Program — Group-based parenting program, 9 weeks delivered in a community setting
  Arms: Parents and Tots Together Program
Behavioral: Supervision for Safety — group-based safety intervention for parents
  Arms: Control

SUMMARY:
This formative research shows that parents of preschool-aged children are enthusiastic about learning general parenting skills, such as discipline strategies, but that they are less interested in information on child nutrition and physical activity needs. To capitalize on this enthusiasm, Dr. Haines developed Parents and Tots Together (PTT), an intervention that embeds strategies to improve children's nutrition and activity behaviours within an existing general skills parenting program. Results from the investigators feasibility trial with 16 Boston-area parents show that PTT is feasible for implementation and is extremely well-received by parents. Results are also encouraging with respect to changing parent feeding behaviours and children's nutrition and activity behaviours. What is not known is whether this program is feasible and contextually appropriate for Canadian families. Thus, the next step in this research program, and the overall goal of this study, is to assess Parents and Tots Together (PTT), a family-based intervention to prevent obesity among children 3 to 5 years of age, within the Canadian context.

To achieve this goal, the investigators will conduct a pilot trial of the PTT program with 60 families recruited through Ontario Early Years Centres (OEYC). The investigators will randomize 30 families to the 3-month PTT intervention and 30 to a control condition.

The investigators primary objective is to implement and test the feasibility and acceptability of PTT among families with preschool children so appropriate revisions can be made to adapt it to a Canadian context. The investigators secondary objective is to compare the following outcomes among intervention versus control participants:

1. Parent weight-related behaviours (i.e., parent physical activity, intake of sugar-sweetened beverages, and television/video viewing, as well as responsiveness to child satiety cues).
2. General parenting behaviours (i.e., use of positive discipline strategies).
3. Child weight-related behaviours (i.e., sleep duration, physical activity, intake of sugar-sweetened beverages, television/video viewing).
4. Nutritional risk score based on a screening tool for preschoolers.
5. Child change in body mass index (BMI), standardized to age and gender.

ELIGIBILITY:
Inclusion Criteria:

* We will consider eligible all parents who have a child age 2-5 years.

Exclusion Criteria:

* We will exclude: 1) any families who plan to move out of the area during the 9-month study period; and 2) children with severe health conditions that would prohibit them from participating in study activities.

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 28 (Actual)
Dates: Start 2013-07; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Child change in body mass index (BMI), standardized to age and gender. | baseline, 6 month follow-up

SECONDARY OUTCOMES:
Change in child sleep duration | baseline, 6-month follow-up
Change in child physical activity | baseline, 6-month follow-up
Change in child intake of sugar-sweetened beverages | baseline, 6-month follow-up
Change in child Television/video viewing | baseline, 6-months
Change in parent feeding behaviours | baseline, 6-months

CONTACTS AND LOCATIONS:
Overall Officials: Jess Haines, Principal Investigator — University of Guelph
Locations (1):
- University of Guelph, Guelph, Ontario, Canada